CLINICAL TRIAL: NCT02907476
Title: The Treatment of Depression With Yoga and Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Partners HealthCare (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-34681; 5R01AT007483-05 (NIH)
Record Dates: First submitted 2016-06-02; First posted 2016-09-20 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Depression; Major Depressive Disorder; PTSD; Anxiety
Keywords: Vagal-gamma amino-butyric acid (GABA); Yoga; Walking
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — Yoga; Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iyengar Yoga (Experimental): Twelve-week Iyengar Yoga protocol with two 90-minute classes per week and three 30-minute homework assignments. Classes consist of approximately 60-minutes of yoga postures, 10-minutes of rest and transition, and 20-minutes of Coherent Breathing at 5 breaths per minute. Homework consist of 15-minutes of yoga postures and 15-minutes of Coherent Breathing. Coherent Breathing is CD guided. Yoga classes are taught by certified Iyengar Yoga instructors.
  Interventions: Behavioral: Iyengar Yoga
- Walking (Active Comparator): Twelve-week walking intervention will consist of two 60-minute group-walking sessions per week and three 15-minute homework walking sessions at 2.5 miles per hour on flat surface. Walking classes are conducted by research staff.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Iyengar Yoga
  Other Names: Yoga
  Arms: Iyengar Yoga
Behavioral: Walking
  Arms: Walking

SUMMARY:
This randomized controlled trial is designed to test the Vagal-gamma amino-butyric acid (GABA) Hypothesis that one of the mechanisms by which yoga-based practices improve mood and decrease anxiety is by correcting an autonomic system (ANS) imbalance with too much activity in the sympathetic nervous system (SNS) and too little activity in the parasympathetic nervous system (PNS). This imbalance is associated with under activity in the GABA system. It is hypothesized that yoga-based practices increase activity in the PNS by increasing respiratory sinus arrhythmia (RSA), which is associated with increased activity in the GABA system and decreased depressive and anxiety symptoms.

DETAILED DESCRIPTION:
Subjects with Major Depressive Disorder (MDD) will be randomized into two treatment groups, a yoga group (YG) and a walking group (WG). After screening and Scan 1, each subject will be randomized to a 12-week yoga or walking intervention consisting of two group sessions and three homework sessions a week.The primary dependent variable will be brain gamma amino-butyric acid (GABA) levels measured using magnetic resonance spectroscopy (MRS) in two regions of interest (ROI)s: the thalamus and the anterior cingulate. GABA levels will be measured three times: Scan 1 prior to randomization, Scan 2 after the 12-week intervention, and immediately after Scan 2, subjects will participate in either the yoga intervention or walking intervention, followed immediately by Scan 3. The secondary dependent variable will be changes in depressive symptoms, mood and anxiety measured by valid and reliable psychological instruments obtained before each scan and at screening, week-4, week-8 and week-12. The third dependent variable will be respiratory sinus arrhythmia (RSA) a component of heart rate variability (HRV) that is an accurately index of vagal influences on the heart. RSA will be measured scan 1, pre and post an intervention session depending on group assignment at week 4, 8 and 12 evaluations, pre and post the yoga or walking intervention between Scan 2 and 3.

Aim 1: To complete 22 subjects in the yoga group and 22 subjects in the walking group for a total of 44 subjects with Major Depressive Disorder (MDD). Completion is defined at a baseline evaluation, a week-4 or week-8 evaluation and a week-12 evaluation with usable thalamic data for Scans 1, 2 and 3.

Aim 2. To measure changes in GABA levels over time using a mixed linear model analogue of repeated measures analysis-of-variance with independent groups in regional GABA levels in MDD subjects assigned to yoga and walking interventions.

Aim 3. To assess changes in psychological measurements and regional GABA levels over the course of the interventions using linear regression.

Aim 4. To assess changes in PNS using Respiratory Sinus Arrhythmia (RSA) over the course of the study using linear regression.

Aim 5. To assess changes in PNS, RSA and regional GABA levels over the course of the study using linear regression.

ELIGIBILITY:
Inclusion Criteria:

* Subject is fluent in English.
* Subject understands the risks and benefits of the study as listed in the Post Consent Quiz.
* Females agree to use an acceptable form of birth control.
* Female had a negative pregnancy test or serum progesterone <= 0.30 ng/ml consistent with the non-luteal phase of the cycle prior to Scan 1.
* Subject meets criteria for Diagnosis of Major Depressive Disorder on the SCID.
* Subject had BDI-II score of at least 14 during screening.
* Subjects who are prescribed a stable dose of antidepressants at least three months with no anticipated changes in their medications for the course of the study (i.e. 3 months after enrollment).
* Subject who have been in a stable form of psychotherapy for three months with no anticipated changes in their psychotherapy for the course of the study (i.e. 3 months after enrollment).
* Subject had given contact information.
* Subject weighs up to 300 lbs at the discretion of the PI.
* Subject has completed all required screening instruments and evaluations.

Exclusion Criteria:

* Subject has a history of psychosis.
* Subject has a history of bipolar illness.
* Subject has a history of suicidal ideation with intent in the last year according to the Columbia Suicide Safety Rating (C-SSR) scale.
* Subject has a history of suicide attempt with attempt to injure in the last year according to the C-SSR.
* Subject who wishes to be treated for MDD with a new treatment during the study such as pharmacotherapy, or somatic therapy or psychotherapy.
* Subject has a contraindication to magnetic resonance evaluation (e.g. pregnancy, a cardiac pacemaker, ferrous implant including shrapnel, or intrauterine devices (IUDs) with copper, claustrophobia that would prevent scanning, some tattoos with black ink on the head including permanent eyeliner).
* Subject has a current mind-body practice (e.g., Tai Chi, Qigong, breathing practices, meditation) defined as more than 6 one-hour sessions in the last 6 months.
* Subject has a current prayer practice > 2 hours a week (prayer group does not count, only prayer practice).
* Subject participates in physical exercise >5 hours/week that is equivalent to or greater than 6 metabolic equivalents (METs) in intensity.
* Subject has been treated with mood stabilizers in the last three months (e.g., Topiramate, Valproic Acid, or Lithium).
* Subject has been treated with medications known to influence the GABA system in the last three months (e.g., anti-anxiety agents such as benzodiazepines, some sleeping aids such as Ambien, or sedative hypnotics).
* Subject uses nicotine regularly in the last three months.
* Subject has a neurologic condition that would in the opinion of the PI would affect the results of the magnetic resonance spectroscopy (MRS) scans.
* Subject has a medical condition that could compromise subject safety or the integrity of the study.
* Subject has a history of having more than 5 alcoholic drinks on 3 or more occasions in the prior three months.
* Subject in the opinion of the PI would not be expected to complete the study including scheduling related issues, whose safety would be jeopardized by participation or who would jeopardize the study protocol.
* Subject has an Axis-I diagnosis, other than depression that in the opinion of the PI would interfere with the subject's participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Brain gamma amino-butyric acid (GABA) levels (change will be measured) | GABA will be measured three times: 1) during screening (scan 1), 2) within 5 weeks after the 12-week intervention (scan 2), 3) immediately following scan 2, but after a yoga or walking session (scan 3).
  Change in GABA levels will be measured using magnetic resonance spectroscopy (MRS) in two regions of interest (ROI)s: the thalamus and the anterior cingulate.

SECONDARY OUTCOMES:
Beck Depression Index Inventory (BDI-II) | Week-12
  The BDI-II is the primary mood scale outcome measure. It is a self-administered scale used to assess symptoms of depression.
Spielberger State-Trait Anxiety Inventory (STAI) | Week-12
  self-administered scale designed for serial assessment of state and trait anxiety.
Exercise-Induced feeling Inventory (EIFI) | Week-12
  Self-administered instrument used to assess feelings states associated with physical activity.
Pittsburgh Sleep Quality Index (PSQI) | Week-12
  Self-administered instrument used to assess sleep quality.
Positivity Self Test (PST) | Week-12.
  Self-administered instrument used to measure positive and negative feelings.
Columbia Suicide Safety Rating (C-SSR) | Week-12
  Clinician-administered instrument to assess suicide risk.
PTSD Check List - Civilian (PCL-C) | Week-12
  Self-Administered measure of PTSD symptoms.
Patient Health Questionnaire 9 (PHQ-9) | Week-12
  Self-Administered instrument used to measure depressive symptoms.

OTHER OUTCOMES:
Heart rate variability (HRV) will be measured by respiratory sinus arrhythmia (RSA), which is an index of vagal influences on the heart. ECG data will be collected to measure RSA using a GGP Biolog IBI monitor (UFI, Morro Bay, CA). | Week-12
  ECG data will be collected using three leads with 6 minutes at rest, three minutes of stepping, followed by six minutes of recovery. post a yoga or walking session, week 12 pre and post a yoga or walking session, and pre and post imaging session 2 (within 3 three weeks of week 12).

CONTACTS AND LOCATIONS:
Overall Officials: Chris C Streeter, MD, Principal Investigator — Boston University
Locations (1):
- Solomon Carter Fuller Building, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is a Data Safety Monitoring Plan that includes Independent Monitors with expertise in the areas of Clinical Care, Imaging and Statistics.